CLINICAL TRIAL: NCT05914272
Title: Association of Osmotic Drugs With Clinical Outcomes in Acute Large Hemispheric Infarction: a Prospective, Multicenter, Observational Cohort Study
Brief Title: Association of Osmotic Drugs With Clinical Outcomes in Acute Large Hemispheric Infarction
Status: Not yet recruiting | Type: Observational
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Collaborators: The Second Hospital University of South China (Other); The Affiliated Hospital of Inner Mongolia Medical University (Other); Second Affiliated Hospital of Wenzhou Medical University (Other); Second Affiliated Hospital of Guangxi Medical University (Other); Fujian Medical University Union Hospital (Other); Huizhou Municipal Central Hospital (Other); Haikou People's Hospital (Other); Kashgar 1st People's Hospital (Other); Ganzhou City People's Hospital (Other); Guangzhou Medical University (Other); Dongguan People's Hospital (Other Government); The First Affiliated Hospital of Hunan University of Traditional Chinese Medicine (Other); Hainan Traditional Chinese Medicine Hospital (Unknown); Hainan People's Hospital (Other); Sinopharm North Hospital (Unknown); Huadu District People's Hospital of Guangzhou (Other); Guangdong Provincial Hospital of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: NFEC-2023-039
Record Dates: First submitted 2023-04-26; First posted 2023-06-22 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Stroke
Keywords: Stroke; large hemispheric infarction; osmotic drugs
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- trement group: Patient has used osmotic drugs within 72 hours of admission.
  Interventions: Drug: Osmotic drugs
- control group: Patient has not used osmotic drugs within 72 hours of admission.
  Interventions: Drug: Osmotic drugs

INTERVENTIONS:
Drug: Osmotic drugs — Patients had used osmotic drugs within 72 hours of admission.

SUMMARY:
Stroke remains the second leading cause of death worldwide, with 2%-8% of these being large hemispheric infarction (LHI) with an occupying effect and the worst prognosis. Even with medical and surgical treatment, the mortality of LHI with cerebral edema is as high as 20% to 30%. Current guidelines recommend supportive supervision, osmotic drugs, and decompressive hemicraniectomy (DHC) for the treatment of LHI, but not all patients with LHI are suitable for DHC, and not all of them can afford the high cost of DHC. In the real-world, the use of osmotic drugs is more common than DHC. The guideline recommends using mannitol or hypertonic saline to reduce cerebral edema and tissue displacement in patients with cerebral edema. Mannitol is the most widely used and longest-standing osmotic drug, and since 1965, hypertonic saline has been used to treat intracranial hypertension. Most of the previous studies compare the efficacy of DHC over medical therapy or compare the efficacy of mannitol with hypertonic saline, but there is an absence of clinical data on whether osmotic drug therapy can improve the clinical prognosis of patients with large hemispheric infarction at 90 days or even longer. Therefore, the purpose of this study was to investigate the association between the osmotic drug and clinical outcomes in large hemispheric infarction, with the aim of informing clinical decisions.

DETAILED DESCRIPTION:
Diagnostic criteria for large hemispheric infarction (LHI): CT within 6 hours of onset showing hypointense areas > 1/3 of the middle cerebral artery territory, or hypointense areas > 50% of the middle cerebral artery territory within 6 hours to 72h of onset. LHI is strongly associated with severe cerebral edema, which can occur to varying degrees cerebral edema within hours or days of LHI. In recent years, endovascular treatment has significantly improved the revascularization of patients with large vessel occlusive cerebral infarction and reduced the incidence of malignant progression and mortality in patients with acute LHI, but many patients still suffer from malignant brain edema (MBE), which leads to the worsening of the disease.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Within 72 hours of onset of the stroke
3. Meets the diagnostic criteria for acute ischaemic stroke in the "Chinese Guidelines for the Diagnosis and Treatment of Acute Ischemic Stroke 2018"
4. Meeting the diagnostic criteria for massive cerebral infarction in the "Guidelines for the Surgical Treatment of Massive Cerebral Infarction": CT within 6 hours of onset showing hypointense areas > 1/3 of the middle cerebral artery territory, or > 50% of the middle cerebral artery territory within 6 hours to 72 hours of onset;
5. The patient consented and signed an informed consent form.

Exclusion Criteria:

1. Women who are pregnant or breastfeeding;
2. in combination with other serious comorbidities resulting in a life expectancy of less than 3 months
3. Those who are allergic or intolerant to osmotic drugs;
4. Those who have participated in other interventional clinical studies (which affecting the observation of outcomes in this cohort);
5. Those with a previous history of stroke and significant residual neurological disability (mRS ≥ 2 points)
6. Those who, in the judgment of the investigator, are not suitable for participation in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acute large hemispheric infarction: CT within 6 hours of onset showing hypointense areas > 1/3 of the middle cerebral artery territory, or > 50% of the middle cerebral artery territory within 6 hours to 72 hours of onset.
Sampling Method: Non-Probability Sample
Enrollment: 2592 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
90-day mortality | 90 days after onset
  Mortality within 90 days after onset in patients with large hemispheric infarction who were eligible for inclusion criteria
Incidence of acute renal impairment | one year after onset
  Incidence of acute renal impairment after onset in patients with large hemispheric infarction who were eligible for inclusion criteria

SECONDARY OUTCOMES:
90-day mRS | 90 days after onset
  Modified Rankin Scale score within 90 days after onset in patients with large hemispheric infarction who were eligible for inclusion criteria
90-day mRS score change | 90 days after onset
  Modified Rankin Scale score change within 90 days after onset in patients with large hemispheric infarction who were eligible for inclusion criteria
one year mRS | 1 year after onset
  Modified Rankin Scale score within 1 year after onset in patients with large hemispheric infarction who were eligible for inclusion criteria
Incidence of early neurological deterioration | 30 days after onset
  Incidence of early neurological deterioration within 30 days after onset in patients with large hemispheric infarction who were eligible for inclusion criteria
Incidence of malignant cerebral edema | 1 year after onset
  Incidence of malignant cerebral edema within 1 year after onset in patients with large hemispheric infarction who were eligible for inclusion criteria
Clinical correction rate of brain herniation before decompressive hemicraniectomy | Up to 3 days
  Clinical correction rate of brain herniation before decompressive hemicraniectomy
Incidence of need for decompressive hemicraniectomy | up to 24 hours
  Incidence of need for decompressive hemicraniectomy after onset
The actual incidence of decompressive hemicraniectomy | up to 24 hours
  The actual incidence of decompressive hemicraniectomy after onset
Incidence of Symptomatic intracranial hemorrhage | up to 24 hours
  Incidence of Symptomatic intracranial hemorrhage within 1 year after onset in patients with large hemispheric infarction who were eligible for inclusion criteria
Incidence of drug-related adverse events | up to 24 hours
  Incidence of adverse events due to drugs within 1 year after the onset of large hemispheric infarction in patients who met the inclusion criteria

CONTACTS AND LOCATIONS:
Overall Officials: Suyue Pan, Principal Investigator — Department of Neurology, Nanfang Hospital, Southern Medical University
Locations (19):
- China (19):
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - Dongguan donghua hospital, Dongguan, Guangdong
  - Dongguan People's Hospital, Dongguan, Guangdong
  - Guangdong Provincial Hospital of Traditional Chinese Medicine, Guangzhou, Guangdong
  - Huadu District People's Hospital of Guangzhou, Guangzhou, Guangdong
  - The Fourth Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Heyuan people's Hospital, Heyuan, Guangdong
  - Huizhou Municipal Central Hospital, Huizhou, Guangdong
  - Haikou People's Hospital, Haikou, Hainan
  - Hainan People's Hospital, Haikou, Hainan
  - Hainan Traditional Chinese Medicine Hospital, Haikou, Hainan
  - The First Hospital of Changsha, Changsha, Hunan
  - The Second Hospital University of South China, Hengyang, Hunan
  - Yueyang People's Hospital, Yueyang, Hunan
  - Sinopharm North Hospital, Baotou, Inner Mongolia
  - The Affiliated Hospital of Inner Mongolia Medical University, Hohhot, Inner Mongolia
  - Ganzhou City People's Hospital, Ganzhou, Jiangxi
  - Kashgar 1st People's Hospital, Kashgar, Xinjiang
  - Second Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang